CLINICAL TRIAL: NCT04699097
Title: Azitromycin Use in COVID-19 Positive Pediatric Patients; Effect on Ventricle Repolarization
Brief Title: The Effect of Azithromycin Use on Conduction System of Heart in COVID-19 Positive Children
Status: Completed | Type: Observational
Sponsor: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, süleyman sunkak, Principal Investigator, Kayseri City Hospital
Other Study IDs: 139
Record Dates: First submitted 2020-12-31; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Azithromycin Adverse Reaction; Covid19; Long QT Syndrome
MeSH Terms: conditions — COVID-19; Long QT Syndrome | interventions — Azithromycin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- azytromycin: children who recieved azithromycin due to COVID 19 infection
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — 250 mg tablet, 5 ml / 200 mg 30 ml suspension

SUMMARY:
Azithromycin (AZ) is used in the pediatric group in COVID-19 diseas. It has been reported to cause prolongation in the QT interval in adult age group. The aim of this study is to evaluate the effect of AZ on ventricular repolarization in COVID-19 positive pediatric patients.

METHOD The study was conducted prospectively in July-August 2020. COVID-19 pediatric patients who received AZ treatment were included in the study. ECG was obtained before treatment and on the 1st, 3rd and 5th days after the treatment. Measurements were made with Image J program®. QTmax, QTmin, Tp-emax, Tp-emin intervals were measured. QTcmax, QTcmin, Tp-ecmax, Tp-ecmin, QTcd, Tp-ecd, and QTc / Tp-ec ratios were calculated with Bazett formula.

DETAILED DESCRIPTION:
The study was prospectively conducted between June 2020 and August 2020. Children hospitalized in Kayseri City Hospital Pediatric Infection Clinic for coronavirus disease and receiving oral AZ treatment were included in the study. Approval was obtained from the local ethics committee. Written informed consent was obtained from the patients and their families. AZ treatment was given as oral 10 mg / kg (maximum 500 mg) on Day 1, followed by 5 mg / kg (maximum 250 mg) on Days 2-5 once a daily. A 12-lead ECG was obtained before the treatment and on the 1st, 3rd and 5th days of the treatment. Patients who did not have at least one ECG before and after the treatment and whose QT and Tp-Te intervals could not be calculated due to excessively parasitic ECG were not included in the study.

ECG was obtained with a GE Mac 2000® device with a paper speed of 25 mm / sec, 10 mv / mm amplitude standard. ECGs were scanned with a scanner and transferred to the computer as JPEG format. QT, Tp-Te intervals were measured by a pediatric cardiologist using ImageJ® program.

Intervals between two consecutive R waves were defined as RR interval. QT interval was defined as the interval from the beginning of the QRS complex to the end of the T wave.

The end of the T wave was defined as intersection of the terminal limb of the T wave with the isoelectric baseline. The longest and the shortest QT intervals across 12 leads were defined as the maximum QT (QTmax) and the minimum QT (QTmin) intervals, respectively. They were corrected according to heart rate by using the Bazett Formula and defined as corrected QTmax (QTmaxc) and corrected QTmin (QTminc), respectively. Bazett formula was preferred to provide uniformity and enable comparison with other studies [Bazett: QTc = QT/(RR)1/2]. QTc dispersion (QTcd) was defined as the difference between QTmaxc and QTminc.

For the T-wave peak to T-wave end interval (Tp-e) measurement, time interval between peak of T wave, ie the time point in which T wave had highest amplitude and end of T wave which also was defined as the crossing point of T wave and isoelectric line was noted as a function of time. Tp-e was also corrected according to heart rate and referred as Tp-ec. The longest and the shortest Tp-e intervals were defined as the maximum Tp-e (Tp-emax) and the minimum Tp-e (Tp-emin) intervals, respectively. Tp-e dispersion (Tp-ed) was defined as the difference between Tp-emax and Tp-emin. Tp-e/QT and Tp-ec/QTc ratios were calculated as maximum and minimum seperately.13 STATISTICAL ANALYSIS The normality of distribution of the ECG measurements and ratios were determined with Kolmogorov-Smirnov test. Descriptive statistics are expressed as mean ± standard deviation (SD) for continuous variables and proportion for categorical variables. Friedman test was used to evaluate repetitive ECG measurements before and after treatment days. P value < 0.05 was considered as statistically significant. All statistical analyses were carried out with the Statistical Package for Social Science for Windows version 22.0 (SPSS Inc., Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

* PCR positive COVID-19 patients
* Age<18 yearts
* Minimum 3 days oral Azithromycin therapy
* At least one ECG before and after treatment

Exclusion Criteria:

* parasitic ECG
* not having at least 1 ECG before or after treatment
* taking drugs other than hydroxychloroquine to prolong the QT interval

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children who recieved oral azithromycin therapy due to COVID 19 infection
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Effect of azitromycin on ventricle repolarization | Before treatment-5th day of treatment
  In the superficial ECG, the QTc, Tp-Tec intervals and Tp-Tec / QTc ratios represent ventricular repolarization. QTc measurement above 0.45 sec is a risk factor for malignant arrhythmia. The significant increase in these intervals and rates compared to previous measurements indicates an increased risk of malignant arrhythmia.

CONTACTS AND LOCATIONS:
Locations (1):
- Süleyman Sunkak, Kayseri, In the USA Or Canada, Please Select..., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
share after 3 months

REFERENCES:
- [Background] McMullan BJ, Mostaghim M. Prescribing azithromycin. Aust Prescr. 2015 Jun;38(3):87-9. doi: 10.18773/austprescr.2015.030. Epub 2015 Jun 1. PMID 26648627
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- [Background] Schwartz RA, Suskind RM. Azithromycin and COVID-19: Prompt early use at first signs of this infection in adults and children, an approach worthy of consideration. Dermatol Ther. 2020 Jul;33(4):e13785. doi: 10.1111/dth.13785. Epub 2020 Jul 12. PMID 32510734
- [Background] Dogan U, Yavas G, Tekinalp M, Yavas C, Ata OY, Ozdemir K. Evaluation of the acute effect of palonosetron on transmural dispersion of myocardial repolarization. Eur Rev Med Pharmacol Sci. 2012 Apr;16(4):462-8. PMID 22696873